CLINICAL TRIAL: NCT03718234
Title: Interval Bolus Delivery of Subcutaneous Hydrocortisone Via Infusion Pump in Children With Congenital Adrenal Hyperplasia
Brief Title: Subcutaneous Hydrocortisone Children With Congenital Adrenal Hyperplasia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEDS-2018-26475; FD-R-6100 (Other Grant/Funding Number: FDA Office of Orphan Products Development)
Record Dates: First submitted 2018-10-11; First posted 2018-10-24 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Congenital Adrenal Hyperplasia; Hyperplasia; Adrenal Hyperplasia; Congenital Disorders; Adrenocortical Hyperfunction; Disorders of Sex Development; Urogenital Abnormalities; Genetic Diseases, Inborn; Steroid Metabolic Diseases, Inborn; Adrenal Gland Disease; Hydrocortisone
Keywords: adrenal gland diseases; cortisol succinate; hydrocortisone; hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Hyperplasia; Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Adrenocortical Hyperfunction; Disorders of Sex Development; Urogenital Abnormalities; Genetic Diseases, Inborn; Steroid Metabolism, Inborn Errors; Adrenal Gland Diseases

STUDY DESIGN:
Intervention Model Description: This is a a single arm non-randomized crossover study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subcutaneous Hydrocortisone via Infusion Pump (Experimental): This is a single arm study. Upon enrollment each participant was admitted for a 24-hr PKPD profile of cortisol, 17OHP and A4 concentrations while on standard oral hydrocortisone therapy (admission 1, week 1). Participant continued on stable oral HC for six weeks. On admission 2, week 7, participant was admitted SQHC pump placement and a safety check was performed to verify absorption of HC was adequate. This consisted of an identical 24-hr PKPD design as used in admission 1. The participants returned to their standard oral HC dosing for 2 weeks while the PKPD profiles from the SQHC pump were being evaluated. The SQHC pump was placed at week 9 and then sent home on the pump. .After 6 weeks of SQHC pump treatment (admission 3, week 14) the participants were admitted and the same 24-hour PKPD design as admissions 1 and 2 profiles was conducted. The subjects were then discharged on their standard oral HC therapy and were followed for an additional 6 weeks
  Interventions: Drug: Subcutaneous hydrocortisone

INTERVENTIONS:
Drug: Subcutaneous hydrocortisone — Pulsatile subcutaneous hydrocortisone administered in 8 doses per day via SQ infusion pump for 6 weeks
  Other Names: Hydrocortisone delivered via subcutaneous pump

SUMMARY:
This is an open-label, non-randomized, single arm proof-of concept feasibility trial comparing standard oral hydrocortisone (HC) treatment with a six-week intervention of interval bolus delivery (pulsatile) of subcutaneous (SQ) HC via infusion pump in children with congenital adrenal hyperplasia (CAH). Eight children, ages 4-18 yrs, will have 24-hr pharmacokinetic and pharmacodynamic (PKPD) profiles of cortisol, 17- hydroxyprogesterone (17OHP) and androstenedione (A4) concentrations while on standard oral hydrocortisone therapy (admission 1, week 1); during a safety check using a subcutaneous hydrocortisone pump (admission 2, week 7); and after 6 weeks of SQHC pump treatment (admission 3, week 14). A pharmacokinetic and pharmacodynamic analysis will be used to compare cortisol, 17OHP and A4 exposures between standard oral HC therapy (week 1) with SQHC pump treatment (week 14). Funding Source - FDA OOPD

ELIGIBILITY:
Inclusion Criteria:

* Children 4 - 18 years of age.
* Classic congenital adrenal hyperplasia (CAH) as confirmed by hormonal and molecular testing.
* Patients who have been on the same HC dosing regimen for 1 month

Exclusion Criteria:

* Patients with non-classic CAH.
* Patients on:

  * Dexamethasone
  * Prednisone, or
  * inhaled steroids.
* Patients with body surface areas under 1m2 or over 2m2
* Non-English speaking patients

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyriaki Sarafoglou, MD, Principal Investigator — University of Minnesota
Locations (1):
- Prism Clinical Research, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramirez Alcantara J, Halper A. Adrenal insufficiency updates in children. Curr Opin Endocrinol Diabetes Obes. 2021 Feb 1;28(1):75-81. doi: 10.1097/MED.0000000000000591. PMID 33278125

RESULTS

PARTICIPANT FLOW:
Groups:
- Subcutaneous Hydrocortisone Via Infusion Pump: Patients will receive a subcutaneous injection of hydrocortisone (HC). Each patient's total daily dose (TDD) of oral tablet hydrocortisone to determine the doses to be delivered of the study drug. The 24-hr schedule and percentage of the TDD of HC will be as follows: approximately 60% of the TDD of HC will be delivered in 3 equal pulses at 0300, 0600 and 0900. Another 35% will be delivered in 3 equal pulses at 1200, 1500 and 1800 and the remaining 5% at 2100 and 2400.
  Subcutaneous hydrocortisone: Patients will be monitored and receive an interval bolus SQHC dosing regimen that more closely mimics cortisol, 17OHP and D4A circadian and ultradian rhythms than conventional oral HC dosing.
Period: Overall Study
Arm/Group | Subcutaneous Hydrocortisone Via Infusion Pump
Started | 11
Completed | 8
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Subcutaneous Hydrocortisone Via Infusion Pump
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cortisol Exposure
Description: 24-hour area under the curve (AUC) following oral hydrocortisone dosing (admission 1).
Time Frame: Week 1
Measure: Mean (Standard Error); unit: hr*mcg/dL
Arm/Group | Subcutaneous Hydrocortisone Via Infusion Pump
Number analyzed (Participants) | 8
hr*mcg/dL | 110 (9.96)

2. Primary Outcome: Cortisol Exposure
Description: The 24-hour cortisol area-under-the curve (AUC) while on the interval bolus delivery (pulsatile) of SQHC (admission 3)
Time Frame: Week 14
Measure: Mean (Standard Error); unit: hr*mcg/dL
Arm/Group | Subcutaneous Hydrocortisone Via Infusion Pump
Number analyzed (Participants) | 8
hr*mcg/dL | 118 (9.10)

3. Primary Outcome: 17-OHP Exposure
Description: 24-hour area under the curve (AUC) following oral hydrocortisone dosing (admission 1).
Time Frame: Week 1
Measure: Mean (Standard Error); unit: hr*ng/dL
Arm/Group | Subcutaneous Hydrocortisone Via Infusion Pump
Number analyzed (Participants) | 8
hr*ng/dL | 46700 (19200)

4. Primary Outcome: 17-OHP Exposure
Description: The 24-hour cortisol area-under-the curve (AUC) while on the interval bolus delivery (pulsatile) of SQHC (admission 3)
Time Frame: Week 14
Measure: Mean (Standard Error); unit: hr*ng/dL
Arm/Group | Subcutaneous Hydrocortisone Via Infusion Pump
Number analyzed (Participants) | 8
hr*ng/dL | 26900 (16200)

5. Primary Outcome: Androstenedione (A4) Exposure
Description: 24-hour area under the curve (AUC) following oral hydrocortisone dosing (admission 1).
Time Frame: Week 1
Measure: Mean (Standard Error); unit: hr*ng/dL
Arm/Group | Subcutaneous Hydrocortisone Via Infusion Pump
Number analyzed (Participants) | 8
hr*ng/dL | 3350 (2410)

6. Primary Outcome: Androstenedione (A4) Exposure
Description: The 24-hour cortisol area-under-the curve (AUC) while on the interval bolus delivery (pulsatile) of SQHC (admission 3)
Time Frame: Week 14
Measure: Mean (Standard Error); unit: hr*ng/dL
Arm/Group | Subcutaneous Hydrocortisone Via Infusion Pump
Number analyzed (Participants) | 8
hr*ng/dL | 1420 (968)

ADVERSE EVENTS:
Time Frame: 20 weeks
Groups:
- Standard Glucocorticoid Therapy: Subjects in this arm will continue on standard oral hydrocortisone therapy
  Standard glucocorticoid therapy: Subjects in this arm will continue on standard oral hydrocortisone therapy
Arm/Group | Subcutaneous Hydrocortisone Via Infusion Pump | Standard Glucocorticoid Therapy
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 9/11 | 9/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subcutaneous Hydrocortisone Via Infusion Pump (N=11) | Standard Glucocorticoid Therapy (N=11)
Stinging/Burning sensation (General disorders) | 8 (11) | 8 (11)
Erythema (General disorders) | 4 (4) | 4 (4)
Itching (General disorders) | 5 (6) | 5 (6)
Skin rash (General disorders) | 1 (1) | 1 (1)
Excoriation (General disorders) | 2 (2) | 2 (2)
Hives (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 2 (4) | 2 (4)
Headache (General disorders) | 1 (1) | 1 (1)
Nasal congestion (General disorders) | 1 (1) | 1 (1)
covid (General disorders) | 1 (1) | 1 (1)
Heartburn (General disorders) | 1 (2) | 1 (2)
Ear infection (General disorders) | 1 (1) | 1 (1)
Streptococcal pharyngitis (General disorders) | 1 (1) | 1 (1)
Respiratory virus (RSV) (General disorders) | 1 (1) | 1 (1)
stomach ache (General disorders) | 1 (1) | 1 (1)
vasovagal syndrome (General disorders) | 1 (2) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT03718234/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/34/NCT03718234/ICF_001.pdf